CLINICAL TRIAL: NCT07074951
Title: Effectiveness of Immunosuppression Combined With Tonsillectomy in Caucasian Patients With High-risk IgA-nephropathy (the Pragmatic Study)
Brief Title: Tonsillectomy and Immunosuppression in Caucasian Patients With High-risk IgA-nephropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director for science RM Gorbacheva Institute, St. Petersburg State Pavlov Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VD285/IgAN/TE+IST
Record Dates: First submitted 2025-06-25; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Primary IgA-nephropathy; High-risk; Caucasians
Keywords: Primary IgA-nephropathy; Corticosteroids; Tonsillectomy; High-risk; Caucasians; Progression; Remission
MeSH Terms: conditions — Glomerulonephritis, IGA; Disease Progression | interventions — Tonsillectomy

STUDY DESIGN:
Intervention Model Description: Experimental group comprises patients, who will receive immunosuppression combined with tonsillectomy (the IST+TE group, n=120).
  Control group includes subjects, fulfilled the same eligibility criteria and underwent only immunosuppression without tonsillectomy in the same time period (the IST group, n=120).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunosuppression combined with tonsillectomy (IST+TE group) (Experimental): Experimental group comprises patients, who will receive immunosuppression combined with tonsillectomy (the IST+TE group, n=120).
  Interventions: Drug: Immunosuppressive treatment; Procedure: Tonsillectomy
- Control group (Active comparator): IST without TE (IST group) (Other): Сontrol group includes subjects with the same eligibility criteria and who will underwent only IST without TE in the same time period.
  Interventions: Drug: Immunosuppressive treatment

INTERVENTIONS:
Drug: Immunosuppressive treatment — Patients will be able to receive the corticosteroid (CS) monotherapy or CS in combination with other immunosuppressive drugs (e.g. cyclophosphamide, mycophenolic acid) by a decision of treating physician.
  CS treatment will start with intravenous or oral induction. In the first case, methylprednisolone will be administered intravenously for 1-3 days at the dosage of 500-1000 mg. Oral prednisolone will be initiated at a dose of 0.5 to 1.0 mg/kg body weight, not exceeded 60 mg/day (week 1) with a rapid decrease by 5 mg each subsequent week until a maintenance dose of 5 mg/day will be reached. Patients will receive maintenance dose for 6 to 12 months.
Procedure: Tonsillectomy — Tonsillectomy will be done in accordance with local clinical practice. TE has to be performed no earlier than 12 months before and no later than 12 months after the initiation of IST.
  Arms: Immunosuppression combined with tonsillectomy (IST+TE group)

SUMMARY:
The open-label prospective non-randomised controlled aims to assess the efficacy of the combination of immunosupression (IST) and tonsillectomy (TE) in Caucasian patients at high risk of the IgA-nephropathy.

ELIGIBILITY:
Inclusion Criteria:

Primary IgA-nephropathy (IgAN) patients with:

1. DP >1 g with haematuria (>5 RBC/HPF)
2. DP <1 g with haematuria AND probability of starting dialysis within 5 years >11% (estimated by the International risk-prediction tool in IgAN) AND at least one of the following histologic changes: at least one of the following histologic changes: mesangial proliferation, endocapillary hypercellularity, cellular crescents

Exclusion Criteria:

1. Age <18 or >75 years;
2. eGFR ≤20 ml/min/1.73m2
3. Patients with mild renal lesions (M0, E0, S0, T0, C0), minor urinary findings, DP <1.0 g
4. Contraindications to IST or TE
5. Patients with any co-existing kidney disease
6. Patients with secondary IgAN (Schoenlein-Henoch purpura, liver cirrhosis, etc.)
7. Patients with diabetes mellitus
8. Any clinically significant acute illness within 60 days prior to kidney biopsy (including infection, aseptic necrosis of any bone, patients with myocardial infarction or cerebrovascular stroke, other conditions that can be exacerbated by corticosteroids
9. Incomplete empiric IST administered prior to kidney biopsy
10. Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 240 (Estimated)
Dates: Start 2013-03-10 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2027-12-10 (Estimated)

PRIMARY OUTCOMES:
Progression | From date of inclusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  The composite end-point of disease progression includes: eGFR decline >40% of baseline level, ESKD (defined as long-term eGFR <15 ml/min/1.73m2 for more than 3 months or need of initiation of renal replacement therapy (RRT).
Overall remission (partial or complete remission) | From date of inclusion until the date of first documented overall remission, assessed up to 120 months
  Partial remission (PR) is defined as a decrease in proteinuria by more than 50% in cases with baseline daily proteinuria (DP) <3.5 g, and in those with DP ≥3.5 g, as its decrease >50% to level <3.5 g/day in combination with regression of hematuria by at least 70% (in 3 consecutive measurements). Complete remission (CR) is defined as DP <0.5 g/day and the disappearance of hematuria (URBC <5/HPF). Any remission is registered in the absence of eGFR decrease >20% from the baseline.
Time to clinical remission | From date of inclusion until the date of first documented remission, assessed up to 120 months
  Cumulative rate of overall (partial or complete) clinical remission

SECONDARY OUTCOMES:
Partial remission | From date of inclusion until the date of first documented partial remission, assessed up to 120 months
  Partial remission is defined as a decrease in proteinuria by more than 50% in cases with baseline DP <3.5 g, and in those with DP ≥3.5 g, as its decrease >50% to level <3.5 g/day in combination with regression of hematuria by at least 70% (in 3 consecutive measurements)
Complete remission | From date of inclusion until the date of first documented complete remission, assessed up to 120 months
  Complete remission is defined as daily proteinuria (DP) <0.5 g/day and the disappearance of hematuria (URBC <5/HPF). Any remission is registered in the absence of eGFR decrease >20% from the baseline.
Relapses | From date of inclusion until the date of first documented relapse, assessed up to 120 months
  In subjects with CR, relapse is defined as the recurrence of proteinuria >1g/day and haematuria (URBC>5/HPF) and, in those with PR, as the increase in proteinuria and haematuria >50% compared to their levels at the time of remission.
The change in proteinuria | Through study completion, an average of 120 months
  Change from baseline in proteinuria
The change in eGFR | Through study completion, an average of 120 months
  Change from baseline in eGFR by CKD-EPI equation
Adverse events per 100 patient-years | From date of inclusion until the date of first documented AE, assessed up to 120 months
  This rate will be expressed as number of adverse events (AEs) per 100 patient-years of observation in every study group. AE grades are based on the NCI Common Terminology Criteria for Adverse Events version 5.0. Serious adverse events (SAEs) are defined according to FDA recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Dobronravov, Professor, MD, PhD, DMedSci, Principal Investigator — St. Petersburg State Pavlov Medical University; Zinaida Kochoyan, Nephrologist, Study Chair — St. Petersburg State Pavlov Medical University
Locations (2):
- Russia (2):
  - Research Institute of Nephrology (Pavlov Medical University), Saint Petersburg
  - St. Petersburg State Pavlov Medical University, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbour SJ, Coppo R, Zhang H, Liu ZH, Suzuki Y, Matsuzaki K, Katafuchi R, Er L, Espino-Hernandez G, Kim SJ, Reich HN, Feehally J, Cattran DC; International IgA Nephropathy Network. Evaluating a New International Risk-Prediction Tool in IgA Nephropathy. JAMA Intern Med. 2019 Jul 1;179(7):942-952. doi: 10.1001/jamainternmed.2019.0600. PMID 30980653